CLINICAL TRIAL: NCT06767813
Title: Multi-cohort, Open, Phase II Clinical Study of TQB2868 Injection Combined With Arotinib Capsule and Chemotherapy in the First-line Treatment of Pancreatic Neoplasms
Brief Title: Clinical Study of TQB2868 Injection Combined With Anlotinib Capsule and Chemotherapy in the First-line Treatment of Metastatic Pancreatic Neoplasms
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2868-ALTN-II-01
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2868 injection+Gemcitabine injection+ Albumin paclitaxel injection+ Anlotinib capsules (Experimental): Treatment period:
  TQB2868 injection combined with Gemcitabine injection and Albumin paclitaxel injection, 28 days as a treatment cycle.
  Oral administration of Anlotinib capsules tablets once a day, for 2 weeks followed by a 1 week untreated recovery phase.
  Maintenance period:
  TQB2868 injection combined with Gemcitabine injection, 21 days as a treatment cycle.
  Oral administration of Anlotinib capsules tablets once a day, for 2 weeks followed by a 1 week untreated recovery phase.
  Interventions: Drug: TQB2868 injection; Drug: Gemcitabine injection; Drug: Albumin paclitaxel injection; Drug: Anlotinib capsules
- TQB2868 injection+Gemcitabine injection +Albumin paclitaxel injection (Experimental): Treatment period TQB2868 injection combined with Gemcitabine injection and Albumin paclitaxel injection, 28 days as a treatment cycle.
  Maintenance period TQB2868 injection combined with Gemcitabine injection, 21 days as a treatment cycle.
  Interventions: Drug: TQB2868 injection; Drug: Gemcitabine injection; Drug: Albumin paclitaxel injection

INTERVENTIONS:
Drug: TQB2868 injection — TQB2868 injection is an anti-PD 1/growth factor (GF)-β Receptor Type II (TGF-βRII) bifunctional fusion protein.
Drug: Gemcitabine injection — Gemcitabine injection
Drug: Albumin paclitaxel injection — Albumin paclitaxel injection
Drug: Anlotinib capsules — Anlotinib capsules
  Arms: TQB2868 injection+Gemcitabine injection+ Albumin paclitaxel injection+ Anlotinib capsules

SUMMARY:
To evaluate the efficacy and safety of TQB2868 injection combined with anlotinib capsule and chemotherapy in treated patients with Pancreatic Neoplasms

ELIGIBILITY:
Inclusion Criteria:

* Subjects must voluntarily participate in the study and sign the informed consent form.
* Aged between 18 and 75 years (inclusive) at the time of signing the informed consent form.
* Diagnosed with pancreatic ductal adenocarcinoma through histological or cytological confirmation.
* Have at least one evaluable metastatic lesion according to RECIST 1.1 criteria;
* No prior systemic anti-tumor therapy (including but not limited to chemotherapy, radiotherapy, targeted therapy, or immunotherapy). Patients who experience disease progression more than 6 months after completing neoadjuvant or adjuvant therapy are eligible.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, with an expected survival of more than 3 months.
* Normal major organ function.
* Patients must use reliable contraception during the study period and for 6 months after the end of the study period; Female participants must have a negative serum or urine pregnancy test within 7 days prior to enrollment and must not be breastfeeding.

Exclusion Criteria:

* Subjects with a history of or concurrent diagnosis of other malignant tumors within the past 5 years.
* Unresolved toxicities from prior treatments exceeding Grade 1 according to Common Terminology Criteria (CTC) AE criteria, excluding alopecia.
* Major surgical procedures, significant traumatic injuries, or unhealed wounds or fractures within 28 days prior to the first dose.
* Any bleeding or hemorrhagic event of ≥ Grade 3 according to CTC AE criteria within 4 weeks prior to the first dose.
* Arterial or venous thrombotic events within 6 months prior to the first dose.
* Active gastric or duodenal ulcers, perforations, persistent positive fecal occult blood tests, ulcerative colitis, or other gastrointestinal bleeding conditions within 6 months prior to the first dose; or other bleeding conditions as assessed by the investigator.
* Hepatitis B virus (HBV)-infected patients unable to adhere to consistent antiviral therapy, or Hepatitis C virus (HCV)-infected patients (positive for HCV Ab or HCV RNA) deemed unstable by the investigator or requiring continued antiviral therapy without consistent adherence.
* History of substance abuse involving psychotropic drugs that cannot be discontinued or presence of psychiatric disorders.
* Symptomatic interstitial lung disease or conditions likely to cause drug-induced lung toxicity or related pneumonitis.
* Presence of any severe and/or uncontrolled diseases.
* Histological or cytological confirmation of other pathological types, such as acinar cell carcinoma, neuroendocrine carcinoma, or pancreatoblastoma.
* Tumors confirmed via imaging (CT or MRI) to have invaded major blood vessels, with the investigator deeming a high likelihood of fatal hemorrhage during the study.
* Tumors confirmed via imaging (CT or MRI) to have invaded the gastrointestinal tract, with a high risk of bleeding based on endoscopy and investigator assessment.
* Known central nervous system metastases and/or carcinomatous meningitis.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage, as assessed by the investigator.
* History of severe allergic reactions to biologic agents or known hypersensitivity to any component of TQB2868 injection.
* Chronic treatment with systemic corticosteroids or other immunosuppressive agents within 28 days prior to the first dose, and continued use of such medications within 2 weeks after the first dose.
* Receipt of live attenuated vaccines within 28 days prior to the first dose or planned administration of live attenuated vaccines during the study.
* Systemic therapy required within 2 years prior to the first dose for any condition. Alternative therapies are not considered systemic therapy.
* Participation in other clinical trials involving anti-tumor drugs within 28 days prior to the first dose.
* Any comorbidities or conditions deemed by the investigator to pose severe risks to the subject's safety or the completion of the study, or any other reasons rendering the subject unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | The evaluation was based on the date of first dose, and efficacy was evaluated every 8 weeks (56±7 days)
  The time between the start of treatment and tumorigenesis (in any aspect) progression or death (due to any cause).
  The evaluation was based on the date of first dose, and efficacy was evaluated every 8 weeks (56±7 days).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | The evaluation was based on the date of first dose, and efficacy was evaluated every 8 weeks (56±7 days)
  The proportion of patients whose tumors have shrunk to a prespecified value and are able to maintain the minimum time limit is the sum of the proportion of complete and partial responses.
Overall survival (OS) | The evaluation was based on the date of first dose, and efficacy was evaluated every 8 weeks (56±7 days)
  Time from the start of treatment to death (due to any cause).
Duration of Response (DOR) | The evaluation was based on the date of first dose, and efficacy was evaluated every 8 weeks (56±7 days)
  The period between the first diagnosis of CR or PR and the discovery of progressive disease (PD).
Disease Control Rate (DCR) | The evaluation was based on the date of first dose, and efficacy was evaluated every 8 weeks (56±7 days)
  The percentage of cases with remission (PR+CR) and stable lesion (SD) after treatment accounted for the number of evaluable cases.
Incidence and severity of adverse events (AEs) | The evaluation was based on the date of first dose, and efficacy was evaluated every 8 weeks (56±7 days)
  The occurrence of all adverse events.
Peak concentration (Cmax) | Day1-7 of cycle1 and cycle 4 : 0 hour pre-dose, 0,1, 2, 4, 8, 24, 48, 72, 144 hours after dose. Cycle1 Day15: 0 hour pre-dose. Day1 of cycle2 and 3 : 0 hour pre-dose. 0 hour after dose, Cycle4 Day15: 0 hour pre-dose. 28days as a cycle.
  Maximum plasma drug concentration.
Transforming growth factor-beta (TGF-β) | Before first dose, 30 minutes after the first dose, pre-dose at Cycle 2 Day 1, pre-dose at the first efficacy assessment, pre-dose at the time of remission at the first efficacy evaluation, and at the time of progression, each cycle is 28 days.
  The relationship between TGF - β content in plasma and anti-tumor efficacy.
Incidence of immunogenicity (ADA) | Cycle1, 2, 4, 8: Before injection. 30 and 90 days after the last dose
  Incidence of immunogenicity (ADA).
Time to maximum blood concentration (Tmax) | Day1-7 of cycle1 and cycle 4 : 0 hour pre-dose, 0,1, 2, 4, 8, 24, 48, 72, 144 hours after dose. Cycle1 Day15: 0 hour pre-dose. Day1 of cycle2 and 3 : 0 hour pre-dose. 0 hour after dose, Cycle4 Day15: 0 hour pre-dose. 28days as a cycle.
  Time to maximum blood concentration.
Area under the time-concentration curve (AUC0-t） | Day1-7 of cycle1 and cycle 4 : 0 hour pre-dose, 0,1, 2, 4, 8, 24, 48, 72, 144 hours after dose. Cycle1 Day15: 0 hour pre-dose. Day1 of cycle2 and 3 : 0 hour pre-dose. 0 hour after dose, Cycle4 Day15: 0 hour pre-dose. 28days as a cycle.
  Area under the time-concentration curve, 0-t hours after administration.
The area under the time-concentration curve ranges from 0 to infinity after administration (AUC0-∞) | Day1-7 of cycle1 and cycle 4 : 0 hour pre-dose, 0,1, 2, 4, 8, 24, 48, 72, 144 hours after dose. Cycle1 Day15: 0 hour pre-dose. Day1 of cycle2 and 3 : 0 hour pre-dose. 0 hour after dose, Cycle4 Day15: 0 hour pre-dose. 28days as a cycle.
  The area under the time-concentration curve ranges from 0 to infinity after administration (AUC0-∞).
Plasma drug half-life (T1/2) | Day1-7 of cycle1 and cycle 4 : 0 hour pre-dose, 0,1, 2, 4, 8, 24, 48, 72, 144 hours after dose. Cycle1 Day15: 0 hour pre-dose. Day1 of cycle2 and 3 : 0 hour pre-dose. 0 hour after dose, Cycle4 Day15: 0 hour pre-dose. 28days as a cycle.
  Plasma drug half-life

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang